CLINICAL TRIAL: NCT07135063
Title: Cranial Nerve Functions in Behçet's Disease and Their Relationship With Clinical Parameters
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MarmaraU-FTR-RHZ-01
Record Dates: First submitted 2025-07-22; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Behcet Disease; Cranial Nerve Disorder
MeSH Terms: conditions — Behcet Syndrome; Cranial Nerve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to find out whether cranial nerves are affected in people with Behçet's Disease (BD), and how this might relate to other disease features. Cranial nerves control important functions such as vision, facial movement, hearing, swallowing, and balance.

The main questions this study will address are:

* Do people with BD have changes in cranial nerve function compared to healthy individuals?
* Are these changes linked to disease duration, symptoms, or lab results?

Participants will:

* Answer questions about their medical history and BD symptoms
* Complete questionnaires on daily function, mood, and autonomic symptoms
* Have a clinical examination of all 12 cranial nerves
* Undergo non-invasive electrical tests to assess nerve function This study will not involve any medications. All procedures will be completed in one visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75
* Diagnosed with BD according to ACR/EULAR 2013 criteria (patient group)
* Healthy with no relevant medical history (control group)

Exclusion Criteria:

* Conditions affecting CN assessment (e.g., facial trauma, surgery, radiotherapy)
* Other rheumatologic or autoimmune diseases
* Psychiatric disorders, alcohol/substance abuse
* Pregnant women
* Use of pacemakers or recent botox to masseter muscle

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Target Population:
  Patient Group: Diagnosed Behçet's patients aged 18-75 years
  Control Group: Age- and gender-matched healthy individuals without neurological, autoimmune, or inflammatory diseases
  Sample Size:
  Minimum 30 Behçet patients
  Minimum 30 healthy controls
  Recruitment:
  Participants will be recruited from Marmara University Pendik Research and Education Hospital. Healthy controls will be volunteers among hospital staff and relatives of patients.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Establish the presence or absence of cranial nerve involvement in BD. | Once: Upon patient inclusion
  Upon patient inclusion EMG and clinical examination is carried out

SECONDARY OUTCOMES:
Investigate relation between disease duration (months) and cranial nerve involvement in BD patients | Once: Upon patient inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Üniversitesi Tıp Fakültesi, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No